CLINICAL TRIAL: NCT01720875
Title: A Phase II Trial of Combination Treatment With Vorinostat, Bortezomib and Dexamethasone in Patients With Relapsed and Relapsed Refractory Multiple Myeloma
Brief Title: Vorinostat, Bortezomib and Dexamethasone in Multiple Myeloma (MUKFour)
Acronym: MUKfour
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Leeds (Other)
Collaborators: Myeloma UK (Other); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HM11/10041; ISRCTN08577602 (Registry Identifier: ISRCTN); 2011-005361-20 (EudraCT Number)
Record Dates: First submitted 2012-10-31; First posted 2012-11-02 (Estimated); Last update posted 2021-08-16 (Actual); Status verified 2021-08

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vorinostat Velcade Dexamethasone (VVD) (Experimental): Up to 8 cycles of VVD followed by vorinostat maintenance until disease progression.
  Cycles 1-8 (21-day cycle)
  * Velcade: 1.3mg/m2 (subcutaneous) on days 1, 4, 8 and 11
  * Dexamethasone: 20 mg (PO) on days 1, 2, 4, 5, 8, 9, 11 and 12
  * Vorinostat: 400mg (PO) on days 1-4, 8-11, 15-18 Maintenance (28-day cycle)
  * Vorinostat: 400mg PO on 1-4 and 15-18
  Interventions: Drug: Vorinostat Velcade Dexamethasone

INTERVENTIONS:
Drug: Vorinostat Velcade Dexamethasone
  Other Names: Bortezomib (velcade)

SUMMARY:
Bortezomib is an established treatment in multiple myeloma; it is common practice in the UK to administer bortezomib with dexamethasone. This practice is based on data that supports improved response rates with this combination.

Recent trial data indicates that the addition of vorinostat to bortezomib treatment overcomes treatment resistance to bortezomib. As such this current trial is designed to investigate the efficacy, safety and tolerability of combination treatment with vorinostat, bortezomib and dexamethasone in patients with relapsed and relapsed refractory myeloma.

A comparison of this Phase II trial with the pivotal Phase III trial conducted by MSD (using the labelled bortezomib indication without dexamethasone) will address the impact of dexamethasone in regards to tolerability and additional efficacy in myeloma patients.

ELIGIBILITY:
Inclusion Criteria:

* Able to give informed consent - Aged 18 years or over
* Participants with relapsed myeloma who have received 1-3 prior lines of treatment and now require further treatment
* ECOG Performance Status ≤ 2
* Required laboratory values within 14 days of registration:

  * Absolute neutrophil count ≥1.0 x 10^9/L.
  * Platelet count ≥75x10^9/L.
  * Haemoglobin > 9 g/dL.
  * Bilirubin ≤1.5 x upper limit of normal
  * ALT and / or AST ≤2.5 x upper limit of normal
  * Serum creatinine ≤ 2.0 x upper limit of normal
  * Corrected calcium ≤ 2.8 mmol/L
* Life expectancy of at least 3 months
* Female participants of child-bearing potential must have a negative pregnancy test at baseline and agree to use dual methods of contraception for the duration of the study and must continue to do so for 3 months after the end of treatment. Male participants must agree to use a barrier method of contraception for the duration of the study if sexually active with a female of child-bearing potential and must continue to do so for 3 months after the end of treatment
* Participant is able to swallow capsules and is able to take or tolerate oral medications on a continuous basis.

Exclusion Criteria:

* Previous anti-tumour therapies, including prior experimental agents or approved anti-tumour small molecules and biologics, within 28 days before the start of protocol treatment. Steroid therapy to stop rapid relapse during this period is permitted, but must be stopped 7 days prior to study drug administration.
* Prior HDAC inhibitor treatment.
* Previous or concurrent active malignancies (<12 months post end of treatment) at other sites with the exception of appropriately treated localised epithelial skin or cervical cancer.
* Participants considered to be refractory to prior bortezomib treatment or unable to tolerate treatment with bortezomib.
* Peripheral neuropathy of ≥ grade 2 severity
* Participants who have received growth factor support or platelet support within 14 days prior to registration
* Participants with uncontrolled concurrent illness or circumstances that could limit compliance with the study.
* Patients with significant cardiovascular or pulmonary disease
* Active symptomatic fungal, bacterial, and/or viral infection including known active HIV or known viral (A, B, or C) hepatitis.
* Pregnant or breast feeding females
* Unable to take corticosteroid therapy at study entry
* Participants with known hypersensitivity to any components of bortezomib, (such as boron, mannitol), vorinostat or dexamethasone.
* Participant has known CNS metastases and/or carcinomatous meningitis.
* Participants with a history of a gastrointestinal surgery or other procedures that might, in the opinion of the Investigator, interfere with the absorption or swallowing of the study drug(s)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2013-08-09 (Actual); Primary Completion 2015-08 (Actual); Study Completion 2018-08-29 (Actual)

PRIMARY OUTCOMES:
Overall response rate to vorinostat, bortezomib and dexamethasone. | up to 24 weeks
  To assess the number and proportion of participants with at least a partial response (PR) or better within 8 cycles of protocol treatment with vorinostat, bortezomib and dexamethasone.

SECONDARY OUTCOMES:
Number of dose reductions during treatment with vorinostat, bortezomib and dexamethasone. | up to 24 weeks
  To assess the dose reduction profile of combination treatment with vorinostat, bortezomib and dexamethasone. The proportion of participants experiencing a dose reduction or terminating treatment early due to toxicity will be assessed.
Overall numbers and rates of adverse events | Up to 18 months
  Safety and toxicity analyses will summarise the overall serious adverse event and adverse events rates including the number and proportion of participants with at least one safety event. SAEs will be additionally presented by the relationship to study treatment, seriousness criteria, event outcome, duration and by MedDRA body system coding.
Progression free survival | Up to 18 months
  A progression-free survival curve will be calculated using the Kaplan Meier method and median PFS estimates will be presented
Maximum response to treatment | Up to 24 weeks
  The overall number and proportion of participants in each response category within 8 cycles of treatment and overall across all treatment including the maintenance phase
Time to maximum response | Up to 18 months
  The time to maximum response will be calculated from the date of registration to the date of maximum response. Participant's who progress and do not achieve a maximum response will be censored at the time of progression. Median time to maximum response will be presented.

OTHER OUTCOMES:
Matched pairs analysis | Up to 24 months
  A matched pairs analysis will be carried out looking at overall response, PFS, dose reductions and toxicity in participants treated with vorinostat in combination with bortezomib and dexamethasone (VVD) in this current study compared to participants randomised to the bortezomib/vorinostat (VV) arm in the pivotal MSD phase III study.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Jenner, Principal Investigator — University Hospital of Southampton
Locations (2):
- United Kingdom (2):
  - Nottingham University Hospital, Nottingham, Nottinghamshire
  - University Hospital Southampton, Southampton

REFERENCES:
- [Result] Brown S, Pawlyn C, Tillotson AL, Sherratt D, Flanagan L, Low E, Morgan GJ, Williams C, Kaiser M, Davies FE, Jenner MW; Myeloma UK Early Phase Clinical Trial Network. Bortezomib, Vorinostat, and Dexamethasone Combination Therapy in Relapsed Myeloma: Results of the Phase 2 MUK four Trial. Clin Lymphoma Myeloma Leuk. 2021 Mar;21(3):154-161.e3. doi: 10.1016/j.clml.2020.11.019. Epub 2020 Dec 3. PMID 33478922